CLINICAL TRIAL: NCT04099927
Title: A Phase I, Open-label Clinical Study on Safety and Pharmacokinetics of SHR0410 Injection for Multiple Administration in Hemodialysis Patients
Brief Title: A Study of SHR4010 in Patients With Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR0410-102
Record Dates: First submitted 2019-08-28; First posted 2019-09-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2020-05

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: SHR0410 monotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR0410 (Experimental): Experimental: SHR0410 dose escalation.
  Interventions: Drug: SHR0410

INTERVENTIONS:
Drug: SHR0410 — SHR0410 monotherapy,given intravenously
  Other Names: KOR agonist

SUMMARY:
The study is being conducted to evaluate the safety and pharmacokinetics of SHR0410 in patients with hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study procedures, the risks involved and obtain written informed consent before any study related activity;
2. Male or female between the ages of 18 and 65 years, inclusive;
3. A total body weight ≥ 50 kg;
4. End stage of renal disease (ESRD) participants who have been on hemodialysis (including hemodiafiltration) for at least six months and are currently on hemodialysis (including hemodiafiltration) three times a week.
5. Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, throughout the study period and for 28 days following last study drug dosing. Female subjects must be post-menopausal for at least 1 year, permanently sterilized (e.g., tubal occlusion, hysterectomy,bilateral salpingectomy) or, if of childbearing potential, must be willing to use a highly effective method of contraception throughout the study period and for 28 days following last study drug dosing, and enter the trial only after menstruation is confirmed..

Exclusion Criteria:

1. Anticipated to receive a kidney transplant during the study;
2. Known history of allergic reaction to opiates such as hives (Note: side effects related to the use of opioids such as constipation or nausea would not exclude the participants from the study);
3. History of drug abuse in the past;
4. Nicotine test positive;
5. Alcohol breath test was positive;
6. The average daily intake of alcohol in the three months before screening was more than 15 g (15 g alcohol equivalent to 450 ml beer or 150 ml wine or 50 ml low-alcohol liquor).
7. Could not obey the unified dietary arrangements and avoid taking coffee or tea during the study period;
8. Blood pressure of upper limbs in supine position was : systolic pressure < 110 mmHg, diastolic pressure < 70 mmHg or systolic pressure > 180 mmHg, diastolic pressure > 110 mmHg at screening or pre-dosing after confirmation in a repeat test;
9. New York Heart Function Classification (NYHA) > III in the screening stage, or abnormal electrocardiogram with clinical significance judged by researchers in the screening stage , including QTcF > 480ms;
10. Screening alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase > 1.5 × ULN, or total bilirubin> 1.5 × ULN.
11. Positive at screening for human immunodeficiency virus (HIV) antibody, Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody.
12. Undergone major surgery within 3 months prior to screening.
13. Total blood loss ≥ 200 ml within 30 days prior to screening, excluding female bleeding during physiological period.
14. Blood human chorionic gonadotropin (hCG) test was positive.
15. Opioids were used within a week before screening, or opioids other than research drugs could not be avoided during the study period.
16. Previous participation in this trial, as defined by signing informed consent form;
17. Participation defined as administration of investigational drugs in another clinical trial (including trial with medical devices) 3 months before screening, or currently participating in another clinical trial (including medical device trials);
18. Any other medical or psychological condition, which in the opinion of the Investigator, might create undue risk to the participant or interfere with the participant's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-28 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | Pre-dose to Day13

SECONDARY OUTCOMES:
Assessment of PK parameter-Area under drug-time curve (AUC0-t) | Pre-dose to Day 6
Assessment of PK parameter-Area under drug-time curve (AUC0-∝) | Pre-dose to Day 6
Assessment of PK parameter-peak time (Tmax) | Pre-dose to Day 6
Assessment of PK parameter-peak concentration (Cmax) | Pre-dose to Day 6
Assessment of PK parameter-half-life (t1/2) | Pre-dose to Day 6
Assessment of PK parameter-pparent clearance rate (CL) | Pre-dose to Day 6
Assessment of PK parameter-apparent distribution volume (Vz) | Pre-dose to Day 6
Pharmacokinetic-The ratio of AUC0-t after the first and last administration. | Pre-dose to Day 6
The renal clearance rate of SHR0410 in urine after each administration. | Pre-dose to Day 6
The cumulative excretion rate of SHR0410 in urine after each administration. | Pre-dose to Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Zou, Study Director — Jiangsu HengRui Medicine Co., Ltd.
Locations (1):
- Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu, China